CLINICAL TRIAL: NCT01664949
Title: A Study to Compare the Safety and Efficacy of A New Eye Drop Formulation With OPTIVE™ in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11002X-001; 2012-002238-35 (EudraCT Number)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carboxymethylcellulose Based Eye Drop Formulation A (Experimental): Carboxymethylcellulose Based Eye Drop Formulation A 1-2 drops in each eye as needed at least 2 times daily for 90 days.
  Interventions: Drug: Carboxymethylcellulose Based Eye Drop Formulation A
- OPTIVE™ (Active Comparator): Carboxymethylcellulose Based Preservative-Free Lubricant Eye Drops (OPTIVE™) 1-2 drops in each eye as needed at least 2 times daily for 90 days.
  Interventions: Drug: Carboxymethylcellulose Based Preservative-Free Lubricant Eye Drops

INTERVENTIONS:
Drug: Carboxymethylcellulose Based Eye Drop Formulation A — Carboxymethylcellulose Based Eye Drop Formulation A 1-2 drops in each eye as needed at least 2 times daily for 90 days.
  Arms: Carboxymethylcellulose Based Eye Drop Formulation A
Drug: Carboxymethylcellulose Based Preservative-Free Lubricant Eye Drops — Carboxymethylcellulose Based Preservative-Free Lubricant Eye Drops (OPTIVE™) 1-2 drops in each eye as needed at least 2 times daily for 90 days.
  Other Names: REFRESH OPTIVE™; OPTAVA™
  Arms: OPTIVE™

SUMMARY:
This study will evaluate the safety and efficacy of a carboxymethylcellulose based eye drop formulation compared with carboxymethylcellulose based preservative-free lubricant eye drops (OPTIVE™) in subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Have used artificial tears for dry eye

Exclusion Criteria:

* Start date of over the counter, herbal, prescription or nutritional supplements that may affect dry eye or vision within 3 months prior to study start or an anticipated change in dosage during the study
* History of eye surgery or trauma in the 6 months prior to study start
* Current use or use within 2 weeks of study start, of topical eye medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (12):
- Randwick, New South Wales, Australia
- Leuven, Belgium
- France (2):
  - Marseille
  - Tours
- Freiburg im Breisgau, Germany
- Italy (2):
  - Padua
  - Parma
- Moscow, Russia
- Spain (2):
  - Huelva
  - Valencia
- United Kingdom (2):
  - Southampton, Hampshire
  - Great Yarmouth, Norfolk

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | OPTIVE™
Started | 224 | 236
Completed | 200 | 211
Not Completed | 24 | 25
Not completed — Adverse Event | 11 | 12
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Personal Reasons | 3 | 4
Not completed — Protocol Violation | 5 | 5
Not completed — Other Miscellaneous Reasons | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | OPTIVE™ | Total
Number analyzed (Participants) | 224 | 236 | 460
Age, Customized [Number; unit: participants]
  < 30 years | 9 (13.77) | 10 (13.65) | 19
  30 to 40 years | 15 | 15 | 30
  > 40 years | 200 | 211 | 411
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 189 | 371
  Male | 42 | 47 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) Score at Day 90
Description: The OSDI consists of 12 questions to assess visual function, ocular symptoms and environmental triggers related to dry eye. Each of the 12 questions is assessed using a 5-point scale (0=none of the time; 4 = all of the time) which is converted to a total score between 0-100. OSDI total scores of 0-12=normal (best), 13-22= mild ocular surface disease, 23-32 =moderate ocular surface disease, and 33-100=severe ocular surface disease (worst). A negative number change from Baseline indicates improvement.
Time Frame: Baseline, Day 90
Population: Participants from the Per-protocol population, all randomized participants without any significant protocol violations, with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | OPTIVE™
Number analyzed (Participants) | 196 | 198
score on a scale
  Baseline | 41.77 (14.018) | 40.92 (13.310)
  Change from Baseline at Day 90 (n=181,185) | -16.88 (17.496) | -15.97 (16.146)

2. Secondary Outcome: Change From Baseline in Tear Break-up Time (TBUT)
Description: TBUT is the time in seconds for the tear film to visually break up after a complete blink. The average of 3 consecutive observations is reported for each participant. The longer it takes, the more stable the tear film. The eye with the shorter average TBUT at Baseline was used for analysis. A positive number change from Baseline indicates improvement.
Time Frame: Baseline, Day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | OPTIVE™
Number analyzed (Participants) | 196 | 198
seconds
  Baseline | 4.50 (1.868) | 4.44 (1.894)
  Change from Baseline at Day 90 (n=181,185) | 2.69 (5.167) | 2.24 (3.262)

3. Secondary Outcome: Change From Baseline in Corneal Staining
Description: Staining of the cornea following ocular administration of fluorescein dye was graded using a 6-point scale (0=no staining, 5=diffuse staining). The eye with the higher score at Baseline was used for analysis. The higher the grade score, the worse the dry eye severity. A negative number change from Baseline indicates improvement.
Time Frame: Baseline, Day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | OPTIVE™
Number analyzed (Participants) | 196 | 198
score on a scale
  Baseline | 1.5 (0.99) | 1.6 (0.99)
  Change from Baseline at Day 90 (n= 182, 184) | -0.7 (0.88) | -0.9 (0.91)

4. Secondary Outcome: Change From Baseline in Conjunctival Staining
Description: Staining of the conjunctiva following ocular administration of lissamine green dye was graded using a 6-point scale (0=no staining, 5=diffuse staining). Conjunctival staining has 2 zones, nasal and temporal, which are added together to provide the total staining score. The eye with the higher score at Baseline was used for analysis. The higher the grade score, the worse the dry eye severity. A negative number change from Baseline indicates improvement.
Time Frame: Baseline, Day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | OPTIVE™
Number analyzed (Participants) | 196 | 198
score on a scale
  Baseline | 2.8 (1.70) | 3.0 (1.79)
  Change from Baseline at Day 90 (n= 181, 185) | -1.3 (1.57) | -1.4 (1.59)

5. Secondary Outcome: Change From Baseline in the Schirmer Test
Description: The Schirmer's Test measures the rate of the secretion of tears produced by the eye over 5 minutes. The results indicate the presence of dry eye. The eye with the lower value at Baseline was used for Analysis. Normal = greater than or equal to 15 millimeters (mm) of tears, Dry Eye = less than 15 mm of tears.. The smaller the number, the more severe the dry eye. A positive number change from Baseline indicates improvement.
Time Frame: Baseline, Day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/5 minutes
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | OPTIVE™
Number analyzed (Participants) | 196 | 198
mm/5 minutes
  Baseline | 9.29 (6.692) | 8.10 (5.888)
  Change from Baseline at Day 90 (n=172,174) | 1.38 (6.933) | 1.53 (6.253)

ADVERSE EVENTS:
Arm/Group | Carboxymethylcellulose Based Eye Drop Formulation A | OPTIVE™
Serious Adverse Events (participants affected / at risk) | 5/224 | 4/236
Other Adverse Events (participants affected / at risk) | 15/224 | 6/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Carboxymethylcellulose Based Eye Drop Formulation A (N=224) | OPTIVE™ (N=236)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1/47 — Adverse Event male specific.
Appendicitis (Infections and infestations) | 0 | 1
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 | 1
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboxymethylcellulose Based Eye Drop Formulation A (N=224) | OPTIVE™ (N=236)
Eye irritation (Eye disorders) | 15 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.